CLINICAL TRIAL: NCT04796168
Title: Post Operative Ankle Splint Study - Prospective Multi Center Randomized Controlled Trial
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait Institute for Medical Specialization (Other Government)
Collaborators: Kuwait University (Other)
Responsible Party: Principal Investigator, Ali Jarragh, Assistant professor, Kuwait Institute for Medical Specialization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1240/2019
Record Dates: First submitted 2021-03-06; First posted 2021-03-12 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Ankle Fractures; Splints
MeSH Terms: conditions — Ankle Fractures | interventions — Calcium Sulfate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post operative Ankle fractures with splint (Active Comparator): All patient who meet the inclusion criteria of having ankle fracture that rigidly fixed and randomized to receive splint post operative
  Interventions: Procedure: Splinting (plaster of paris)
- post operative Ankle fractures without splint (No Intervention): All patient who meet the inclusion criteria of having ankle fracture that rigidly fixed and randomized to receive NO splint post operative

INTERVENTIONS:
Procedure: Splinting (plaster of paris) — Placing stockinette followed by cotton rolls and 10-12 layer of posterior ankle splint made of plaster of paris
  Arms: post operative Ankle fractures with splint

SUMMARY:
Background: Ankle fractures are some of the most common orthopedic presentations, however, controversy in their management and their post-operative rehabilitation protocols exist. Most displaced ankle fractures treated with anatomical reduction and stable internal fixation to allow early range of motion by allowing rigid fixation and restoration of ankle joint congruence. Post-operative rehabilitation protocols varies between surgeons and institutions with the majority emphasising early rehabilitation protocols. The use of a splint. The rational for splinting ankle fractures after rigid fixation is to decrease pain level, rest the soft tissues and prevent equinus deformity. Up to date there is no scientific research to question the benefit of routine use of splints after rigid fixation of ankle fractures.

Methods: A prospective multi-centre randomised control trial. Approximately fifty patients will be enrolled from 3 hospitals (Adan, Mubarak and Farwaniya hospital) over a 1 year period. The studied sample will be randomised into 2 groups using computerised randomisation software: splint group and no-splint group. The patients will be examined at set intervals for pain, swelling, deep-vein thrombosis and a set of scoring tools. The tools include: visual analogue score (VAS) for pain, Short Form Health Survey (SF-36), American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot score, physical and radiological assessment at 2 weeks, 3 months, 6 months and 1 year intervals. Statistical Package for the Social Sciences program (SPSS) will be used for statistical analysis

Results/outcomes: Functional scores, symptoms and signs, complications, radio-graphic and clinical follow up will be recorded.

DETAILED DESCRIPTION:
Overview

The mainstay of unstable ankle fractures is surgical in nature, however controversy and an unclear consensus exists regarding post-operative rehabilitation; is a splint necessary or not? Splinting the ankle post-op is traditionally used to reduce pain and limit motion. However, the evidence is unclear and benefits are not well established. Further, splinting the ankle in the traditional back-slab is accompanied by complications including; pressure sores, skin irritation and deep-vein thrombosis.

There is incomplete evidence supporting early commencement of weight-bearing and the use of a detachable type of immobilization to allow exercise during the immobilization period after surgical fixation(1). It is also noteworthy that its believed that because of the potential increased risk of adverse events, the patient's compliance with the use of a removable type of immobilisation to enable controlled exercise is essential(1). To date there is lacking scientific research to question the benefit of routine use of splints after rigid fixation of ankle fractures. There is little evidence that any specific rehabilitation program improves clinical outcome (2). One study found that active ankle movements in combination with weight bearing facilitate and improve the rehabilitation following operation for an ankle fracture [3]. A systematic review of 38 controlled trials related to the rehabilitation of ankle fractures found that early ambulation post-op may improve ankle range of motion, yet with limited quality evidence [3, 6]. . Early performance of ankle exercises following surgical fixation improved ankle function and mobility, while decreasing pain, but was associated with higher rates of adverse events (e.g. surgical wound complications), although most problems were minor(3). Use of a removable immobilization device was necessary for this approach. It could be plausible that determent and harm to the patient is being done in the form of dermatological adverse effects of splints if there is in fact no benefit to their use. There is a clear need to define whether or not a splint is needed for the sake of patient safety and comfort postoperatively.

Research Question/Hypothesis What are the benefits and risks of splinting ankle fractures post-op. The investigators believe that there is no considerable benefit to splinting ankle fractures after fixation, in fact, splinting may even result in stiffness, cast-associated complications and reduced patient satisfaction.

Objectives and aims

Overall Objective To critically assess the benefits of splints after rigid fixation of ankle fractures.

Specific Aims

1- To assess the level of pain between the splint and no-splint groups. 2- To compare the range of motion between the splint and no-splint groups. Secondary objectives

1. To assess patient satisfaction between the splint and no-splint groups.
2. To assess other complications and radiological finding differences between the splint and no-splint groups.
3. To check the difference in time-to-union between the splint and no-splint groups.

BACKGROUND AND SIGNIFICANCE

Ankle fractures

Over five million ankle injuries occur each year in the United States alone, and the incidence of these fractures is approximately 187 fractures per 100,000 people each year (4). This figure has been increasing, most probably because of the exponential growth of the population and the growing amount of people practising sports(4). Cigarette smoking and a high body mass index have been associated with ankle fractures(5, 6). Ankle fractures can be categorised into stable and unstable fractures. Isolated malleolar fractures are usually stable if they are not displaced but, care should be taken with fractures of the medial malleolus. Disturbance of nearby structures often occurs in association with these fractures, and they sometimes appear to be isolated injuries at first. Bimalleolar Fractures, which is fracture of both the lateral and medial malleoli, are generally unstable. Trimalleolar fractures are unstable and typically occur with injuries of greater force. These are bimalleolar fractures with a fracture of the posterior malleolus.

Fracture stability determines treatment. Emergent conditions, such as an open fracture or neurovascular impairment, necessitate surgical consultation and treatment. Fracture dislocations must be reduced to avoid serious complications, such as avascular necrosis. After emergency situations are excluded, the fracture should be evaluated more closely, with focus on any malalignment or instability, to determine proper management. Standard treatment for stable ankle is Immobilization in a cast (CI) for approximately six weeks but, new evidence is growing and supporting that shorter periods of casting allows a similar level of healing with less risk of complications. A randomized trial of 247 adults with stable fractures of the lateral malleolus, 3 week long immobilization in a short-leg walking cast or rigid ankle orthosis reduced the short-term loss of ankle mobility and the risk for deep vein thrombosis as compared with care, without compromising fracture healing(4). Confirmation of these results is needed, but 3 weeks of immobilization may be a reasonable approach in healthy adults with uncomplicated fractures. Unstable ankle fractures are treated surgically.

Research design and methods

Overview

The PASS Trial is going to be a 1-2 year long randomised control trial where a qualified team of doctors will administer a questionnaire, take clinical examination results, and assign patients to treatment groups of splint and non-splint post-surgical repair. Range of motion will be evaluated with a Goniometer and information will be gathered in a standardized manner. Patients aged 18-65 taken from Adan, Mubarak, and Farwaniya hospitals will be consented and randomly assigned to a treatment group after which they will be followed periodically at their designated follow up appointments, which are at 2 weeks, 3 months, 6 months and 1 year. Patients will be collected over the duration of 2 years until a quota of 50-75 participants is achieved. Only isolated A.O 44 ankle fractures requiring surgical fixation will be included in the study. Pathological fractures, polytrauma patients and open fractures will be excluded.

Strengths and weaknesses of the study

Study Design

This study is a double blinded Randomized Control Trial to eliminate as much bias as possible. All Principle investigators who measured the results are near equal in terms of experience and education. Methods of gathering and collecting data as well as tools to do so were standardized. Our study will utilize multivariate regression models and intention to treat analysis. The study covers the major trauma centres in Kuwait providing adequate representation of the population. Recall bias is minimized due to close proximity of questioning and the event.

Potential Limitations Patient compliance to treatment arms is the main potential issue of our study. The extent of non-compliance was measured through questionnaire. There is a lack of literature on this subject, which results in deficient comparison with other populations around the globe and in the region.

Public health significance

On the Individual Level The Patients as individuals will feel liberated as they may no longer consider themselves disabled and diseased while they are not wearing a split providing physiological relief. This benefit could even translate to earlier return to work and benefit society. Individuals will no longer be inconvenienced by being required to wear a splint.

On The Global Level It is in the interest of public health care systems to conduct this trial because there is a possibility that the costs of splints provide by the hospitals will be cut and put to better use. Such a trial could impact public health policy because it can provide good evidence to change the current standards of care. This study may also reveal associations that are possibly good targets for public health intervention. This is especially important in our country as there is a locally observed predisposition to injury for hard labour and construction workers, so there it is necessity to see if there is an association between current working conditions and likeliness of injury.

ELIGIBILITY:
Inclusion Criteria:

* A.O 44 ankle fractures requiring surgical fixation (uni or bimalleolar with /without syndesmotic injury)

Exclusion Criteria:

* pathological fracture
* poly trauma pilon fractures open fractures other associated fractures in same extremity peripheral neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Assessing the change in the level of pain between the splint and no-splint groups | Change in pain from 2 weeks postop to 1 year postop
  Visual analogue scale (0;lowest pain, 10;highest pain)
Assessing the change in ankle swelling from 2 weeks postop to 1 year postop in the splint and no-splint groups | Change in swelling from 2 weeks postop to 1 year postop
  Measuring tape to assess supramalleolar, mid-foot, and mid-calf circumference

SECONDARY OUTCOMES:
Change in the functional scoring system used below | Change in American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scorefrom 2 weeks postop to 1 year postop
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score
Number of participants with; infection, nonunion, deep-vein thrombosis, stiffness, equinus | From 2 weeks postop - 1 year postop
  Rate of infection, nonunion, deep-vein thrombosis, stiffness, equinus

CONTACTS AND LOCATIONS:
Overall Officials: Ali Jarragh, MD, Principal Investigator — Kuwait University
Locations (1):
- Mubarak Al kabeer hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michelson JD. Fractures about the ankle. J Bone Joint Surg Am. 1995 Jan;77(1):142-52. doi: 10.2106/00004623-199501000-00020. No abstract available. PMID 7822349
- [Background] Ahl T, Dalen N, Selvik G. Mobilization after operation of ankle fractures. Good results of early motion and weight bearing. Acta Orthop Scand. 1988 Jun;59(3):302-6. doi: 10.3109/17453678809149368. PMID 3132812
- [Background] Daly PJ, Fitzgerald RH Jr, Melton LJ, Ilstrup DM. Epidemiology of ankle fractures in Rochester, Minnesota. Acta Orthop Scand. 1987 Oct;58(5):539-44. doi: 10.3109/17453678709146395. PMID 3425285
- [Background] Valtola A, Honkanen R, Kroger H, Tuppurainen M, Saarikoski S, Alhava E. Lifestyle and other factors predict ankle fractures in perimenopausal women: a population-based prospective cohort study. Bone. 2002 Jan;30(1):238-42. doi: 10.1016/s8756-3282(01)00649-4. PMID 11792591
- [Background] Honkanen R, Tuppurainen M, Kroger H, Alhava E, Saarikoski S. Relationships between risk factors and fractures differ by type of fracture: a population-based study of 12,192 perimenopausal women. Osteoporos Int. 1998;8(1):25-31. doi: 10.1007/s001980050044. PMID 9692074
- [Background] Smeeing DP, Houwert RM, Briet JP, Kelder JC, Segers MJ, Verleisdonk EJ, Leenen LP, Hietbrink F. Weight-bearing and mobilization in the postoperative care of ankle fractures: a systematic review and meta-analysis of randomized controlled trials and cohort studies. PLoS One. 2015 Feb 19;10(2):e0118320. doi: 10.1371/journal.pone.0118320. eCollection 2015. PMID 25695796
- [Result] Lin CW, Donkers NA, Refshauge KM, Beckenkamp PR, Khera K, Moseley AM. Rehabilitation for ankle fractures in adults. Cochrane Database Syst Rev. 2012 Nov 14;11:CD005595. doi: 10.1002/14651858.CD005595.pub3. PMID 23152232